CLINICAL TRIAL: NCT06203249
Title: Microecology and Host Immunity in Patients With Anti-melanoma Differentiation Associated Gene 5 Antibody Positive Dermatomyositis and Interstitial Lung Disease
Brief Title: Microecology and Immunity in Patients With Anti-MDA5 Antibody Positive Dermatomyositis and Interstitial Lung Disease
Status: Recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, wang kaifei, Chinese PLA General Hospital, Chinese PLA General Hospital
Other Study IDs: Microecology and Immunity 1
Record Dates: First submitted 2023-12-28; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Microbiome; Immune Function; Anti-MDA5 Antibody Positive Dermatomyositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — bronchoalveolar lavage specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study was to analyze the relationship between the microbial community, host immunity and the presence or absence of concurrent rapidly progressive interstitial lung disease patients with anti-MDA5 antibody positive dermatomyositis.

DETAILED DESCRIPTION:
Methods: Bronchoalveolar lavage specimens of patients with anti-MDA5 antibody positive dermatomyositis and interstitial lung disease were collected and studied to analyze the relationship between the composition of patients' microecology and the occurrence and development of disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria of dermatomyositis and anti-MDA 5 antibody positive.
* Anti-MDA5 antibody positive DM patients with RPILD meet the diagnostic criteria for RPILD.
* Must have undergone bronchoalveolar lavage.
* Age≥18 years old.
* Patients who signed informed consent forms

Exclusion Criteria:

* Patients who had other connective tissue diseases.
* Patients with ILD or RPILD caused by infection, tumors, drugs, biochemistry and other factors.
* Pregnant or lactating patients.
* The patient also participated in any other clinical trial.
* Disagreement for inclusion in this study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anti-MDA5 antibody positive dermatomyositis patients with or without interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
The relationship between the microbial community and the presence or absence of interstitial lung disease | 6 months
  The relationship between the microbial community and the presence or absence of interstitial lung disease

CONTACTS AND LOCATIONS:
Locations (1):
- PLA, Beijing, Beijing Municipality, China